CLINICAL TRIAL: NCT06711952
Title: German Validation Study of the Subjective Cognitive Decline Questionnaire (SCD-Q) and Its Potential Use in Large Cohorts
Brief Title: German Validation Study of the Subjective Cognitive Decline Questionnaire (SCD-Q)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Medotrax UG (Unknown)
Responsible Party: Principal Investigator, Robert Perneczky, Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 22-1117
Record Dates: First submitted 2023-12-21; First posted 2024-12-02 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Subjective Cognitive Decline
Keywords: Alzheimer's Disease; Subjective Cognitive Decline; German Validation
MeSH Terms: conditions — Alzheimer Disease | interventions — Environmental Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjective Cognitive Decline Questionnaire (SCD-Q) (Other): Participants receive treatment as usual (appointment in the memory clinic, LMU) and will additionally fill out the questionnaires. A digital cognitive test will be performed.
  Interventions: Diagnostic Test: Subjective Cognitive Decline-Questionnaire (SCD-Q); Diagnostic Test: Cognitive Failure Questionnaire (CFQ); Diagnostic Test: biomarkers; Diagnostic Test: Cognitive Tests

INTERVENTIONS:
Diagnostic Test: Subjective Cognitive Decline-Questionnaire (SCD-Q) — The SCD-Q is an established instrument to quantify self-perceived cognitive decline. In addition to the self-perceived cognitive complaints, a 24 items questionnaire of informants is part of SCD-Q. The self-reported SCD-Q will be included in the standard health questionnaire that all patients of the memory clinic of the LMU Department of Psychiatry and Psychotherapy are required to complete before the examination date. The health questionnaire will be sent per mail. All routine clinical procedures will remain unchanged.
Diagnostic Test: Cognitive Failure Questionnaire (CFQ) — The Cognitive Failure Questionnaire (CFQ) is a questionnaire for measuring self-reported subjective failures in cognition, memory and motor functions in everyday life. The German CFQ consists of 32 items related to everyday possibilities of error, whose frequency in the last six months is to be estimated by means of a five-point rating scale.
Diagnostic Test: biomarkers — Blood plasma and serum samples will be collected by the project staff according to standard operating procedures used at LMU Munich and subsequently processed and measured at the Department of Psychiatry and Psychotherapy to quantify the blood-based biomarkers for AD using Elecsys immunoassays running on a Cobas e402 analyzer.
  Only available clinical and biomarker data will be used (Routine cerebrospinal fluid biomarkers, routine imaging biomarkers).
Diagnostic Test: Cognitive Tests — The investigators plan to examine the patients´ visuospatial performance on site with a digital clock-drawing test, which has been validated in large community-based studies.
  The Functional Activities Questionnaire (FAQ) shall be filled out by an informant. FAQ is a reliable and valid measure of activities of daily living. The results of the routine neuropsychological tests (Consortium to Establish a Registry for AD, Mini-Mental-State Examination) will be used in the analysis.

SUMMARY:
The SCD-Q (Subjective Cognitive Decline-Questionnaire) is an established instrument to quantify self-perceived cognitive decline. Both self- and informant-rated versions of the SCD-Q are available. However, the SCD-Q has not been validated in the German language yet. Hence, the investigators aim to validate the self-reported SCD-Q in a clinical sample in Germany.

DETAILED DESCRIPTION:
The SCD-Q is a well-established screening instrument to quantify perceived subjective cognitive decline. In addition to self-perceived cognitive complaints, a 24-item questionnaire for informants is part of the SCD-Q. It demonstrates high sensitivity and lower specificity for detecting dementia and early cognitive changes associated with dementia. However, the questionnaire has not been translated into German or validated. Plasma biomarkers for amyloid and tau pathology, as well as for neurodegeneration and astrocytic activation, have been developed and show promising sensitivity and specificity for detecting Alzheimer's disease (AD). A relevant proportion of biomarker-positive patients does not convert to mild cognitive impairment or Alzheimer's disease dementia during the disease course. Currently, the predictive value of blood biomarkers remains to be clarified, particularly in conjunction with SCD. This study aims to validate the SCD-Q in German and analyze possible connections with biomarkers and (digital) cognitive tests. Follow-up visits are planned.

ELIGIBILITY:
Inclusion Criteria:

* Medical appointment for dementia diagnostics at the Alzheimer Therapie- und Forschungszentrum
* Provision of signed, written and dated informed consent
* Capacity to give informed consent

Exclusion Criteria:

* dementia in a very advance stage
* Illiteracy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Validation of the SCD-Q in the german language | Baseline
  assessment of its psychometric properties, including reliability, validity, and sensitivity/specificity, when translated into German.(neuropsychological test, neurological and psychiatric examination, MRI and optional lumbar puncture), sensitivity and specifity to identify participants with probable AD, establish cut-off values of the SCD-Q; • Internal consistency of the self-rated SCD-Q (measured by Cronbach's alpha).
  * Test-retest reliability (correlation coefficient between repeated measures at two time points).
  * Construct validity (comparison with related cognitive self-assessment tools or scales).
  * Discriminative ability (sensitivity and specificity for distinguishing between individuals with subjective cognitive decline and those without, using ROC analysis).
  * Linguistic validation process (forward and backward translation, followed by expert review and pilot testing).
combination of SCD-Q and biomarkers | Baseline
  To determine and validate appropriate cut-off values for the self-rated SCD-Q for distinguishing between individuals with and without subjective cognitive decline. • Receiver Operating Characteristic (ROC) analysis to establish sensitivity and specificity of the SCD-Q.
  * Optimal cut-off values derived using Youden's Index to maximize diagnostic performance.
  * Units of Measure: SCD-Q total score (range: 0-100).
Correlation of SCD-Q with digital cognitive tests and a shortened version of SCD-Q | Baseline
  correlation of the SCD-Q with a digital cognitive test and shortened version of the SCD-Q.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Perneczky, Prof. Dr., Principal Investigator — Klinik und Poliklinik für Psychiatrie und Psychotherapie des LMU Klinikums
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie des LMU Klinikums, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No